CLINICAL TRIAL: NCT01657812
Title: A Comparison of Dexmedetomidine and Epidural Anesthesia Under General Anesthesia in Patients Undergoing Gastrectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Yun Li, Head of department of Anesthesiology in the Second Affiliated Hospital of Anhui Medical University, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3869480
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Gastrectomy
Keywords: dexmedetomidine; Epidural Anesthesia; stress response; anesthesia recovery
MeSH Terms: conditions — Fractures, Stress | interventions — Dexmedetomidine; Injections, Epidural

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- dexmedetomidine (Experimental): Drug:dexmedetomidine,dexmedetomidine 1.0μg/kg intravenous injection within 15 minutes before the induction of general anesthesia and followed by Dex 0.4μg/kg/h until 40min before the end of surgery
  Interventions: Drug: dexmedetomidine
- epidural (Active Comparator): Epidural:continuous epidural block (T8-9) 4 mL of 1.6% lidocaine as a test dose and continous infusion of 0.375% ropivacaine(5 mL/h) during the surgery
  Interventions: Drug: dexmedetomidine
- control (Placebo Comparator): Drug: normalsaline

INTERVENTIONS:
Drug: dexmedetomidine — Dexmedetomidine, an alpha 2 agonist provides sedative, anxiolytic, anti-shivering, analgesic, and anaesthetic sparing effect. In addition α2-adrenoceptor agonists reduce central sympathetic outflow and attenuate the stress response associated with surgery.Unlike epidural anaesthesia, dexmedetomidine is easy to administer and no potential for neurological damage.
  Date suggest that the dexmedetomidine reduces the stress response of surgery to the similar extent to epidural anaesthesia when used in conjunction with a standard general anaesthesia for abdominal surgery.
  Other Names: epidural
  Arms: dexmedetomidine; epidural

SUMMARY:
Clinically, combining epidural with general anaesthesia may confer many advantages to patients undergoing major thoracic, abdominal or orthopaedic surgery. Epidural anaesthesia can attenuate sympathetic hyperactivity and the stress response, maintain bowel peristalsis, spare the use of opioids, and facilitate postoperative feeding and physiotherapy. However, establishing epidural anesthesia is not without risks and contraindications, including refusal by the patient, technical failure, unintentional dural puncture, waist and back pain and local anaesthetic toxicity. When neurologic complications do occur, the resulting morbidity and mortality is considerable. Dexmedetomidine is a potent α2-adrenoceptor agonist with an 8 times greater affinity for α2-adrenoceptors than clonidine. This class of agent is known to have sedative, anxiolytic, anti-shivering, analgesic, and anaesthetic sparing effect. In addition α2-adrenoceptor agonists reduce central sympathetic outflow and attenuate the stress response associated with surgery.1 Unlike epidural anaesthesia, dexmedetomidine is easy to administer and no potential for neurological damage. The investigators hypothesize that the dexmedetomidine reduces the stress response of surgery to the similar extent to epidural anaesthesia when used in conjunction with a standard general anaesthesia for abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Consent
* ASA 1-2
* No contraindication to epidural or dexmedetomidine
* First time surgery for current conditions
* Not on chronic pain medications or sedative

Exclusion Criteria:

* .The subject has known significant renal or hepatic disorders determined by medical history, physical examination or laboratory tests

  * The subject has a known or suspected allergy to opioid analgesics or dexmedetomidine
  * The subject has history of. cardiovascular issues which would preclude the use of dexmedetomidine
  * The subject has know central nervous system disease or neurological impairment
  * The subject is an ASA classification of 3 or greater

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-06 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Parameters: Heart rate, blood pressure and ECG ;Parameters on stress response:norepinephrine (NE), epinephrine ( E) | pre-administration of Dex or epidural anesthesia,intubation, 3 min after intubation , immediately after incision, immediately after the initiation of celiac exploration, 1 h after operation,extubation

SECONDARY OUTCOMES:
Anesthetics consumption: propofol and remifentanil consumption | during operation
anesthesia recovery :the time of eye opening, side effects such as nausea, vomiting and post-anaesthetic shivering, VAS, first exhaust time, hospitalization time | up to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ye Zhang, Ph.D, Principal Investigator — The Second Hospital of Anhui Medical University
Locations (1):
- The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

REFERENCES:
- [Background] Kunisawa T, Nagata O, Nagashima M, Mitamura S, Ueno M, Suzuki A, Takahata O, Iwasaki H. Dexmedetomidine suppresses the decrease in blood pressure during anesthetic induction and blunts the cardiovascular response to tracheal intubation. J Clin Anesth. 2009 May;21(3):194-9. doi: 10.1016/j.jclinane.2008.08.015. PMID 19464613